CLINICAL TRIAL: NCT04426968
Title: A Phase II Randomized, Double-blind, Placebo-controlled, Multi-center, Dose-effect Relationship Study of Hepalatide for Injection Combined With Pegylated Interferon in Subjects With Chronic Hepatitis B
Brief Title: A Phase II Study of Hepalatide in Subjects With Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai HEP Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L47-HB-II-02
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2022-12

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hepalatide 2.1mg+Pegylated Interferon (Experimental): Hepalatide 2.1mg s.c., q.d., treatment continued for 24 weeks, follow up 4 weeks.
  PEG-IFNalpha, s.c., q.w.,treatment continued for 48 weeks
  Interventions: Drug: Hepalatide 2.1mg; Drug: Pegylated Interferon
- Hepalatide 4.2mg+Pegylated Interferon (Experimental): Hepalatide 4.2mg s.c., q.d., treatment continued for 24 weeks, follow up 4 weeks.
  PEG-IFNalpha, s.c., q.w.,treatment continued for 48 weeks
  Interventions: Drug: Hepalatide 4.2mg; Drug: Pegylated Interferon
- Hepalatide 6.3mg+Pegylated Interferon (Experimental): Hepalatide 6.3mg s.c., q.d., treatment continued for 24 weeks, follow up 4 weeks.
  PEG-IFNalpha, s.c., q.w.,treatment continued for 48 weeks
  Interventions: Drug: Hepalatide 6.3mg; Drug: Pegylated Interferon
- placebo+Pegylated Interferon (Active Comparator): Hepalatide placebo s.c., q.d., treatment continued for 24 weeks, follow up 4 weeks.
  PEG-IFNalpha, s.c., q.w.,treatment continued for 48 weeks
  Interventions: Drug: placebo 2.1mg; Drug: placebo 4.2mg; Drug: placebo 6.3mg; Drug: Pegylated Interferon

INTERVENTIONS:
Drug: Hepalatide 2.1mg — 2.1 mg/day subcutaneously (s.c.) for 24 week
  Other Names: L47
  Arms: Hepalatide 2.1mg+Pegylated Interferon
Drug: Hepalatide 4.2mg — 4.2mg/day subcutaneously (s.c.) for 24 week
  Other Names: L47
  Arms: Hepalatide 4.2mg+Pegylated Interferon
Drug: Hepalatide 6.3mg — 6.3mg/day subcutaneously (s.c.) for 24 week
  Other Names: L47
  Arms: Hepalatide 6.3mg+Pegylated Interferon
Drug: placebo 2.1mg — 2.1 mg/day subcutaneously (s.c.) for 24 week
  Arms: placebo+Pegylated Interferon
Drug: placebo 4.2mg — 4.2 mg/day subcutaneously (s.c.) for 24 week
  Arms: placebo+Pegylated Interferon
Drug: placebo 6.3mg — 6.3 mg/day subcutaneously (s.c.) for 24 week
  Arms: placebo+Pegylated Interferon
Drug: Pegylated Interferon — 180 ug/week subcutaneously (s.c.) for 28 week
  Other Names: Pegasys

SUMMARY:
A Phase II Randomized, Double-blind, Placebo-controlled, Multi-center, Dose-effect Relationship Study of Hepalatide for Injection Combined with Pegylated Interferon in Subjects with Chronic Hepatitis B

DETAILED DESCRIPTION:
The study is a 4-arm parallel design, randomized, double-blind, placebo-controlled, multicenter, dose-effect relationship, phase II clinical trial. The study is designed to assess efficacy and safety of 3 Doses of hepalatide in Combination with Pegylated Interferon Compared to Pegylated Interferon Alone in patients with Chronic Hepatitis B .Subjects will be randomly assigned to the 2.1mg, 4.2mg, and 6.3mg dose groups , 32 subjects in each group . The subjects in each dose group will be randomly and double-blindly administered the corresponding dose of trial drug or placebo in a ratio of 3:1. The subjects in each dose group who received placebo treatment combine as the placebo group. All subjects will receive Pegylated Interferon treatment for 28 weeks as the basic treatment,trial drug or placebo treatment for 24 weeks continuously , followed by a safety follow-up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 60 years inclusively at the time of signing Informed Consent Form.
2. HBsAg or/and HBV DNA Positive for at least 6 months before Screening.
3. Subjects did not receive interferon treatment and did not receive nucleotide/nucleoside analogue within 6 months
4. HBeAg positive or negative
5. HBV DNA≥20,000 IU/ml (HBeAg positive) or HBV DNA≥2,000 IU/ml (HBeAg negative)
6. 2×ULN ≤ALT≤10×ULN
7. Serum total bilirubin<2×ULN
8. Subjects had no history of decompensated liver disease（Ascites, jaundice, hepatic encephalopathy, varicose hemorrhage）, serious heart disease (including unstable or uncontrolled heart disease within 6 months),serious mental illness (especially depression),organ transplantation .subjects have no uncontrolled epilepsy, mental illness, diabetes and hypertension,no autoimmune disease, immune related extrahepatic manifestations (vasculitis, purpura, nodular arteritis, peripheral neuropathy and glomerulonephritis), thyroid disease, malignant tumor, immunosuppressive therapy; no basic diseases and other serious diseases such as serious infection, retinal disease, heart failure and chronic obstructive pulmonary disease; no alcohol and drug abuse.
9. Subjects must agree to use a highly effective contraception for 2 years , female subjects are not pregnant or breastfeeding
10. Subjects did not donate blood or as clinical trial subjects within 3 months before screening
11. Subjects have good compliance with the protocol
12. Subjects understood and agreed to sign the informed consent form.

Exclusion Criteria:

1. Decompensated liver disease: direct bilirubin > 1.2 × ULN,
2. Prothrombin time > 1.2 × ULN, serum albumin < 35 g / L
3. Severe liver fibrosis or cirrhosis: METAVIR score of liver biopsy is 4 points; or or Child-Pugh score> 7
4. Hemocytopenia: neutrophil < 1 × 10^9 / L, platelet < 50 × 10^9 / L, hemoglobin < 100g / L (female) or hemoglobin < 110g / L (male) points
5. HAV,HCV,HDV,HEV or HIV infection
6. Pegylated interferon therapy is contraindicated
7. Allergic to interferon, Such as severe depression, epilepsy, autoimmune diseases, uncontrolled thyroid dysfunction and so on
8. severe retinopathy or eye disease(Eye diseases due to high blood pressure or diabetes, CMV retinitis, macular degeneration)
9. Positive for anti-HBV Pre-S1 antibody.
10. Hamilton Depression Scale (HAMD, 17 items) score > 17 points
11. Female subjects pregnancy test positive
12. Other laboratories or auxiliary examinations are obviously abnormal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
virological response | 24weeks

SECONDARY OUTCOMES:
HBV DNA down from baseline | 24weeks
  HBV DNA down from baseline log10

OTHER OUTCOMES:
Virological suppression | 24weeks
  HBV DNA <2,000 IU/ml
No response | 24weeks
  HBsAg >20,000 IU/ml and HBV DNA lower than baseline <2log10 IU/ml
Partial virological response | 24weeks
  HBV DNA >20 IU/ml and ≥2log10 IU/ml lower than baseline
HBsAg is down from baseline | 24weeks
  HBsAg is down from baseline log10
HBeAg turned negative | 24weeks
  HBeAg <0.05 index
HBeAg is down from baseline | 24weeks
  HBeAg is down from baseline log10
ALT recurrence | 24weeks
  ALT≤1.25×ULN
Histological response | 24weeks
  Liver tissue inflammatory necrosis score reduced by ≥2 points with no increased liver fibrosis score; liver fibrosis score reduced by ≥1 point

CONTACTS AND LOCATIONS:
Overall Officials: Fusheng Wang, Principal Investigator — The fifth medical center of PLA
Locations (12):
- China (12):
  - The fifth medical center of PLA, Beijing, Beijing Municipality
  - Jilin Hepatobiliary Disease Hospital, Changchun
  - The first hospital of Jilin University, Changchun
  - Chizhou People's Hospital, Chizhou
  - The First Hospital Affiliated to the Army Medical University, Chongqing
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Hospital of Nanjing, Nanjing
  - Qingyuan People's Hospital, Qingyuan
  - Shanghai Tongren Hospital, Shanghai
  - The Sixth People's Hospital of Shenyang, Shenyang
  - Henan Provincial People's Hospital, Zhengzhou
  - Henan Provincial Infectious Disease Hospital, Zhenzhou

IPD SHARING:
Plan to Share IPD: No